CLINICAL TRIAL: NCT03502577
Title: A Phase I Study of B-Cell Maturation Antigen (BCMA)-Specific Chimeric Antigen Receptor T Cells in Combination With JSMD194, a Small Molecule Inhibitor of Gamma Secretase, in Patients With Relapsed or Persistent Multiple Myeloma
Brief Title: BCMA-Specific CAR T-Cells Combined With a Gamma Secretase Inhibitor (JSMD194) to Treat Relapsed or Persistent Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9952; NCI-2018-00514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9952 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9218033 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; crenigacestat; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Chemotherapy, BCMA-specific CAR T-cells, LY3039478) (Experimental): Participants receive fludarabine and cyclophosphamide on days -4 to -2. Participants then receive BCMA-specific CAR T-cells IV over 20-30 minutes on day 0 and LY3039478 PO on days 2, 4, 7, 9, 11, 14, 16, and 18.
  Interventions: Biological: BCMA-specific CAR-expressing T Lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Gamma-Secretase Inhibitor LY3039478; Other: Laboratory Biomarker Analysis; Other: Pharmacokinetic Study

INTERVENTIONS:
Biological: BCMA-specific CAR-expressing T Lymphocytes — Receive CAR T infusion
  Other Names: Anti-BCMA CAR T Cells; Anti-BCMA-CAR-transduced T Cells
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Gamma-Secretase Inhibitor LY3039478 — Given PO
  Other Names: LY 3039478; LY-3039478; LY3039478; JSMD194
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase I trial determines the side effects and best dose of B-cell maturation antigen (BCMA)-chimeric antigen receptor (CAR) T-cells when combined with gamma-secretase inhibitor LY3039478 (JSMD194), cyclophosphamide, and fludarabine in treating participants with multiple myeloma that that has come back or remains despite treatment. Placing genes added in the laboratory into immune T-cells may make the T-cells recognize BCMA, a protein on the surface of cancer cells. JSMD194 may enhance the killing of cancer cells by increasing the BCMA expression on multiple myeloma cells, making the targeted BCMA CAR-T treatment more effective. JSMD194 also decreases the amount of BCMA found in the circulation (called soluble BCMA) that is not bound to the myeloma cells. JSMD194 can therefore reduce the potential for soluble BCMA to act as a decoy. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving BCMA CAR T therapy with JSMD194, cyclophosphamide, and fludarabine may work better in treating participants with relapsed or persistent multiple myeloma.

DETAILED DESCRIPTION:
OUTLINE: This is a dose escalation study of BCMA-specific CAR T-cells.

Participants receive fludarabine and cyclophosphamide on days -4 to -2. Participants then receive BCMA-specific CAR T-cells intravenously (IV) over 20-30 minutes on day 0 and gamma-secretase inhibitor LY3039478 orally (PO) on days 2, 4, 7, 9, 11, 14, 16, and 18. Patients will also receive JSMD194 orally before the fludarabine and cyclophosphamide to evaluate the effect of this drug alone on multiple myeloma cell BCMA levels.

After completion of study treatment, participants are followed up every 6 months for years 1-5 and annually for years 6-15.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score =< 2
* Have measurable disease by International Myeloma Working Group (IMWG) criteria based on one or more of the following findings:

  * Serum monoclonal immunoglobulin (M-protein) >= 1 g/dL
  * Urine M-protein >= 200 mg/24 hour
  * Involved serum free light chain (sFLC) level >= 10 mg/dL with abnormal kappa/lambda ratio
  * Measurable biopsy-proven plasmacytomas (>= 1 lesion that has a single diameter >= 2 cm)
  * Bone marrow plasma cells >= 30%
* Have a diagnosis of multiple myeloma (MM); the MM diagnosis must be confirmed by internal pathology review of a fresh biopsy specimen at the Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance (FHCRC/SCCA)
* Have relapsed or treatment refractory disease with >= 10% CD138+ malignant plasma cells immunohistochemistry (IHC) on BM core biopsy, either:

  * Following autologous stem-cell transplantation (ASCT)
  * Or, if a patient has not yet undergone ASCT, the individual must:

    * Be transplant ineligible, due to age, comorbidity, patient choice, insurance reasons, concerns of rapidly progressive disease, and/or discretion of attending physician and principal investigator and,
    * Demonstrate disease that persists after > 4 cycles of induction therapy and that is double refractory (persistence/progression) after therapy with both a proteasome inhibitor (PI) and immunomodulatory drug (IMiD) administered either in tandem, or in sequence, or demonstrate intolerance to both classes of agents (IMiD and PI); > 4 cycles of therapy are not required for patients with a diagnosis of plasma cell leukemia
* Male and female patients of reproductive potential must be willing to use an effect contraceptive method before, during, and for at least 4 months after the BCMA CAR T cell infusion

Exclusion Criteria:

* History of another primary malignancy that requires intervention beyond surveillance or that has not been in remission for at least 1 year (the following are exempt from the 1-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer, curatively treated superficial bladder cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear)
* Active hepatitis B, hepatitis C at the time of screening
* Patients who are human immunodeficiency virus (HIV) seropositive
* Subjects with uncontrolled active infection
* > 1 hospital admission for infection in prior 6 months
* Presence of acute or chronic graft-versus-host disease (GVHD) unless limited to skin involvement and managed with topical steroid therapy alone
* History of any one of the following cardiovascular conditions within the past 6 months: class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease as determined by the principal investigator (PI) or designee
* History of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis, active central nervous system MM involvement and/or carcinomatous meningitis; subjects with previously treated central nervous systems involvement may participate, provided they are free of disease in the CNS (documented by flow cytometry performed on the cerebrospinal fluid [CSF] within 14 days of enrollment) and have no evidence of new sites of CNS activity
* Pregnant or breastfeeding females
* Allogeneic hematopoietic stem cell transplantation (HSCT) or donor lymphocyte infusion within 90 days of leukapheresis
* Use of any of the following:

  * Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis; physiologic replacement, topical, and inhaled steroids are permitted
  * Cytotoxic chemotherapeutic agents within 1 week of leukapheresis; oral chemotherapeutic agents are allowed if at least 3 half-lives have elapsed prior to leukapheresis
  * Lymphotoxic chemotherapeutic agents within 2 weeks of leukapheresis
  * Experimental agents within 4 weeks of leukapheresis unless progression is documented on therapy and at least 3 half-lives have elapsed prior to leukapheresis
  * Daratumumab (or other anti-CD38 therapy) within 30 days of leukapheresis
* Absolute neutrophil count (ANC) < 1000/mm^3, per PI discretion if cytopenia thought to be related to underlying myeloma
* Hemoglobin (Hgb) < 8 mg/dl, per PI discretion if cytopenia thought to be related to underlying myeloma
* Platelet count < 50,000/mm^3, per PI discretion if cytopenia thought to be related to underlying myeloma
* Active autoimmune disease requiring immunosuppressive therapy
* Creatinine clearance < 20 ml/min
* Significant hepatic dysfunction (serum glutamic-oxaloacetic transaminase [SGOT] > 5 x upper limit of normal; bilirubin > 3.0 mg/dL)
* Forced expiratory volume in one second (FEV1) of < 50% predicted or carbon monoxide diffusing capacity (DLCO) (corrected) < 40% (patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing)
* Anticipated survival of < 3 months
* Contraindication to cyclophosphamide or fludarabine chemotherapy
* Patients with known amyloidosis (AL) subtype amyloidosis
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the investigator; or unwillingness or inability to follow the procedures required in the protocol
* Documented malabsorptive syndromes including enteropathies, gastroenteritis (acute or chronic) or diarrhea (acute or chronic)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of chimeric antigen receptor (CAR) T cells | Up to 28 days following CAR T-cell infusion
  This is defined as the dose associated with a true dose-limiting toxicity (DLT) rate of 25% in each of the cohorts. DLTs are events that occur within the first 28 days following CAR T-cell infusion.
Incidence of general toxicities | Up to 1 year
  This will be measured according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission | Up to 1 year
Progression-free survival | Up to 1 year
Overall survival | Up to 1 year
Duration of persistence of adoptively transferred B-cell maturation antigen (BCMA) CAR T cells | Up to 1 year
Evaluation of the migration of adoptively transferred BCMA CAR T cells | Up to 1 year

OTHER OUTCOMES:
Plasma cell BCMA expression and soluble (s)BCMA levels with LY3039478 administration | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cowan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowan AJ, Pont MJ, Sather BD, Turtle CJ, Till BG, Libby EN 3rd, Coffey DG, Tuazon SA, Wood B, Gooley T, Wu VQ, Voutsinas J, Song X, Shadman M, Gauthier J, Chapuis AG, Milano F, Maloney DG, Riddell SR, Green DJ. gamma-Secretase inhibitor in combination with BCMA chimeric antigen receptor T-cell immunotherapy for individuals with relapsed or refractory multiple myeloma: a phase 1, first-in-human trial. Lancet Oncol. 2023 Jul;24(7):811-822. doi: 10.1016/S1470-2045(23)00246-2. PMID 37414012
- [Derived] Pont MJ, Hill T, Cole GO, Abbott JJ, Kelliher J, Salter AI, Hudecek M, Comstock ML, Rajan A, Patel BKR, Voutsinas JM, Wu Q, Liu L, Cowan AJ, Wood BL, Green DJ, Riddell SR. gamma-Secretase inhibition increases efficacy of BCMA-specific chimeric antigen receptor T cells in multiple myeloma. Blood. 2019 Nov 7;134(19):1585-1597. doi: 10.1182/blood.2019000050. PMID 31558469